CLINICAL TRIAL: NCT01433354
Title: An Open-label Study to Evaluate the Long-term Safety and Tolerability of AFQ056 in Adolescent Patients With Fragile X Syndrome
Brief Title: Long-term, Safety and Tolerability Study of AFQ056 in Adolescent Patients With Fragile X Syndrome (Open-label)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study treatment failed to demonstrate efficacy in target population in two other clinical studies (CAFQ056B2214 and CAFQ056A2212).
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAFQ056B2278; 2011-002379-40 (EudraCT Number)
Record Dates: First submitted 2011-08-31; First posted 2011-09-13 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Martin-Bell Syndrome; Genetic Diseases; X-Linked; Escalante's syndrome
MeSH Terms: conditions — Fragile X Syndrome; Genetic Diseases, Inborn | interventions — mavoglurant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFQ056 Treatment (Experimental): All patients will initiate treatment with AFQ056 at a starting dose of 25 mg b.i.d. The dose will be titrated from 25 mg b.i.d to 50 mg b.i.d., 75 mg b.i.d. and 100 mg b.i.d. at weekly intervals. Dose adjustments (up- and down-titrations) will be permitted as needed to manage any tolerability issues and to ensure that patients reach their highest tolerated dose, not to exceed 100 mg b.i.d.
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056 — The investigational drug, AFQ056, will be provided as hard gelatin capsules. Two different oral dosage strengths,25mg and 100 mg, identical in appearance, will be used.

SUMMARY:
The purpose of this study is to generate long-term safety, tolerability and efficacy data for AFQ056 in eligible adolescent patients with FXS who have participated in the CAFQ056B2214 study, the PK study CAFQ056B2131, or another study of AFQ056 which included FXS patients below 18 years of age provided the patient is at least 12 years of age at the time of entry into the current study.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 patients:
* Must have completed study CAFQ056B2214 or another study of AFQ056 which included FXS patients below 18 years of age within one week of enrollment into the open-label study.
* Has a caregiver or caregivers who spend, on average, at least 6 hours per day with the patient , who is willing to and capable of supervising treatment, providing input into efficacy and safety assessments, and accompanying the patient to study visits.
* Group 2 patients:
* Must meet one of the following conditions:
* Completed Study CAFQ056B2131
* Completed Study CAFQ056B2214 or another study of AFQ056 which included FXS patients below 18 years of age but enrollment into the current study was delayed for more than a week.
* Discontinued prematurely from Study CAFQ056B2214 or another study of AFQ056 which included FXS patients below 18 years of age due to intolerability of the dosage in the patient's assigned treatment group.
* Has a caregiver or caregivers who spend, on average, at least 6 hours per day with the patient , who is willing to and capable of supervising treatment, providing input into efficacy and safety assessments, and accompanying the patient to study visits.

Exclusion Criteria:

* Discontinuation from Study CAFQ056B2214 or CAFQ056B2131 or another study of AFQ056 which included FXS patients below 18 years of age due to safety reasons
* Female patients who are sexually active at any time during the study
* Any advanced, severe or unstable disease
* History and/or presence of schizophrenia, bipolar disease, psychosis, confusional states and/or repeated hallucinations as per DSM-IV criteria
* History of suicidal behavior or considered a high suicidal risk
* History of severe self-injurious behavior
* History of uncontrolled seizure disorder or resistant to therapy within the past 2 years (Patients who are clinically stable under anti-convulsant therapy for the past 2 years are not excluded)
* History of clinically significant allergies requiring hospitalization or non-inhaled corticosteroid therapy (asthma, anaphylaxis, etc.)
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether or not there is evidence of local recurrence or metastases
* Patients who are using (or used within 6 weeks before baseline) digoxin or warfarin
* Using (or used within 6 weeks before baseline) concomitant medications that are potent inhibitors or inducers of CYP3A4
* Using glutamatergic agents (riluzole, memantine, etc.) or lithium within 6 weeks of baseline

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (7):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Nashville, Tennessee
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Glostrup Municipality, Denmark
- Novartis Investigative Site, Bron, France
- Germany (4):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Padua
- Novartis Investigative Site, Rotterdam, Netherlands
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Novartis Investigative Site, Spånga, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Bailey DB Jr, Berry-Kravis E, Wheeler A, Raspa M, Merrien F, Ricart J, Koumaras B, Rosenkranz G, Tomlinson M, von Raison F, Apostol G. Mavoglurant in adolescents with fragile X syndrome: analysis of Clinical Global Impression-Improvement source data from a double-blind therapeutic study followed by an open-label, long-term extension study. J Neurodev Disord. 2016;8:1. doi: 10.1186/s11689-015-9134-5. Epub 2015 Dec 15. PMID 26855682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 centres in 13 countries.
Pre-assignment Details: A total of 120 patients were enrolled, of which 119 received the study medication. Category 1 patients received AFQ056 in the core study and enrolled in the extension within 7 days of the core study; Category 2 included all other patients who were enrolled into the extension study
Groups:
- AFQ056: Participants from a previous AFQ056 study who entered the open-label extension study were administered AFQ056 capsules at a starting dose of 25 milligram (mg) twice daily (bid) and then titrated to 50 mg bid, 75 mg bid and 100 mg bid at weekly intervals.
Period: Overall Study
Arm/Group | AFQ056
Started | 119 (120 enrolled of which 119 were administered drug)
Completed | 0
Not Completed | 119
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Administrative problems | 90
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 17
Not completed — Subject Withdrew Consent | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of the study drug (AFQ056) during the study.
Arm/Group | AFQ056
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events were summarized for the open-label treatment period, where the open-label treatment period is defined based on how AEs were collected and reported according to the manner in which participants entered the current study and which treatment (AFQ056 or placebo) they were receiving in the previous study.
  AEs which were continuing from the core study or that started after the end of core study but prior to first dose of open-label study medication in the extension study for Category 1 participants are shown under 'Prior to Ext. first dose'.
  AEs which started during the open-label treatment period are presented based on the last AFQ056 dose taken on or before the onset date of the AE (25 mg bid; 50 mg bid; 75 mg bid; or 100 mg bid). No efficacy data presented as study was terminated.
Time Frame: Prior to first dose in extension study, Baseline (start of study treatment in extension study) to End of trial
Population: The analysis was performed in the safety set (SS) population, defined as participants who received at least one dose of study medication and had at least one safety assessment occurring after first dose of extension study medication. Here, 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Groups:
- AFQ056: Total
Arm/Group | AFQ056 | Prior to Ext. First Dose | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 75 mg Bid | AFQ056 100 mg Bid
Number analyzed (Participants) | 119 | 31 | 119 | 118 | 116 | 108
participants
  At least one AE | 110 | 10 | 36 | 41 | 44 | 90
  At least one severe AE | 8 | 0 | 1 | 1 | 1 | 5
  Any serious or significant AE | 4 | 0 | 0 | 1 | 0 | 3
  SAEs | 4 | 0 | 0 | 1 | 0 | 3
  Discontinued due to AEs | 6 | 1 | 2 | 2 | 0 | 3
  Discontinued due to SAEs | 1 | 0 | 0 | 0 | 0 | 1
  Discontinued due to non serious AE | 5 | 1 | 2 | 2 | 0 | 2

ADVERSE EVENTS:
Groups:
- Prior to Ext.First Dose: Prior to Ext.first dose
- AFQ056 25 mg Bid: AFQ056 25 mg bid
- AFQ056 50 mg Bid: AFQ056 50 mg bid
- AFQ056 75 mg Bid: AFQ056 75 mg bid
- AFQ056 100 mg Bid: AFQ056 100 mg bid
- Total: Total
Arm/Group | Prior to Ext.First Dose | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 75 mg Bid | AFQ056 100 mg Bid | Total
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/119 | 1/118 | 0/116 | 3/108 | 4/119
Other Adverse Events (participants affected / at risk) | 6/31 | 23/119 | 30/118 | 33/116 | 74/108 | 103/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Ext.First Dose (N=31) | AFQ056 25 mg Bid (N=119) | AFQ056 50 mg Bid (N=118) | AFQ056 75 mg Bid (N=116) | AFQ056 100 mg Bid (N=108) | Total (N=119)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Ext.First Dose (N=31) | AFQ056 25 mg Bid (N=119) | AFQ056 50 mg Bid (N=118) | AFQ056 75 mg Bid (N=116) | AFQ056 100 mg Bid (N=108) | Total (N=119)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 4 | 0 | 5 | 12
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 0 | 8 | 13
Fatigue (General disorders) | 0 | 2 | 2 | 3 | 5 | 11
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 4 | 7
Ear infection (Infections and infestations) | 0 | 2 | 0 | 1 | 5 | 8
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 1 | 5 | 8
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 6 | 8
Nasopharyngitis (Infections and infestations) | 0 | 7 | 3 | 8 | 25 | 35
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 5 | 3 | 9 | 17
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 5 | 7
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 0 | 5
Headache (Nervous system disorders) | 0 | 4 | 1 | 4 | 8 | 15
Psychomotor hyperactivity (Nervous system disorders) | 0 | 2 | 3 | 1 | 3 | 9
Aggression (Psychiatric disorders) | 0 | 3 | 3 | 4 | 12 | 19
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 4 | 6
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 0 | 11 | 15
Initial insomnia (Psychiatric disorders) | 0 | 3 | 2 | 4 | 9 | 18
Insomnia (Psychiatric disorders) | 1 | 4 | 10 | 5 | 12 | 25
Irritability (Psychiatric disorders) | 0 | 3 | 1 | 3 | 9 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4 | 7 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 3 | 6

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate this study prematurely, as the study treatment failed to demonstrate efficacy in target population in two other clinical studies: CAFQ056B2214 (NCT01357239) and CAFQ056A2212 (NCT01253629).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.